CLINICAL TRIAL: NCT04385498
Title: Posttraumatic Stress Disorder Intervention for People With Severe Mental Illness in Low- and Middle-Income Country Primary Care Settings
Brief Title: Primary Care Intervention for PTSD in Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Addis Ababa University (Other)
Responsible Party: Principal Investigator, Lauren Ng, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-001993
Record Dates: First submitted 2020-04-28; First posted 2020-05-13 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: PTSD
Keywords: Post Traumatic Stress Disorder; Severe Mental Illness; psychotherapy; global mental health; Ethiopia
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BREATHE Intervention (Experimental): Five session program, with additional sessions provided based on the individual's learning style and needs. Sessions are designed to be 20 to 30 minutes long, to accommodate the needs of the primary health care centers. Sessions will ideally be conducted once per week, but may be conducted as infrequently as once per month.
  Interventions: Behavioral: BREATHE Intervention
- Waitlist Treatment as Usual (Active Comparator): Typical primary care treatment which will include medication management and follow-up at the health facilities, at at least the same frequency as treatment arm. At the End of the trial participants will be able to receive the BREATHE Ethiopia PTSD treatment
  Interventions: Behavioral: Waitlist Treatment as Usual

INTERVENTIONS:
Behavioral: BREATHE Intervention — 5 session program focusing on breathing retraining, psychoeducation, and positive coping.
  Other Names: BREATHE Ethiopia
  Arms: BREATHE Intervention
Behavioral: Waitlist Treatment as Usual — Typical primary care treatment which will include medication management and follow-up at the health facilities, at at least the same frequency as treatment arm. At the end of the trial Participants will be able to receive the BREATHE Ethiopia treatment.
  Arms: Waitlist Treatment as Usual

SUMMARY:
Mixed methods (qualitative and quantitative) cluster randomized pilot feasibility trial (n=40) to refine the the Brief Relaxation, Education and Trauma Healing (BREATHE) Ethiopia intervention and explore effectiveness and implementation. Fifty patients will be enrolled across the pre-pilot and the pilot to account for potential treatment dropout. Eight health care centers will be randomized to Treatment or Waitlist conditions.

1. Primary outcomes: Change in hypothesized treatment mechanisms: (1) increased knowledge about PTSD; reductions in (2) PTSD-related stigma; (3) trauma-related cognitions; and (4) self-reported arousal; (5) increased use of stress management strategies; and (6) reductions in physiological arousal as measured by increased heart rate variability.
2. Secondary outcomes: Change in symptoms and functional impairment. Reductions in (1) PTSD (2) depression and anxiety symptoms, and (3) functional impairment.
3. Process evaluation: Mixed methods multi-stakeholder process evaluation of the implementation of the intervention as measured by the RE-AIM framework (Reach, Effectiveness, Adoption, Implementation, Maintenance). We will collect qualitative data on Adoption and Implementation (e.g. facilitators and barriers to intervention delivery) and quantitative assessment of patient and provider participation and retention (Reach), satisfaction (Adoption) and fidelity (Implementation).

ELIGIBILITY:
Inclusion Criteria:

1. For all participants: Being 18 years of age or older
2. For all participants: Being able and willing to provide informed consent to participate in the study
3. For all participants: Being able to complete procedures in Amharic or English.
4. For patients: Treatment at a Sodo district primary care clinic for Severe Mental Illness (SMI)
5. For patients: Identified as having:

   1. Experienced a traumatic event,
   2. Associated PTSD symptoms defined as scores on the PTSD Checklist DSM-5 (PCL-5), AND
   3. any associated functional impairment on the WHODAS-2.
6. For health care providers: Providers working at the target health centers who administer, provider care for, or supervise the care of patients with mental health concerns.
7. For caregivers: Being identified by the patient as a close family member or friend whom the patient gives permission to be involved in the study

Exclusion Criteria:

1. Current high risk of suicide as measured by the Composite International Diagnostic Interview (CIDI) Suicide module
2. Inability to participate in the treatment, as determined by the psychiatric nurse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Change in PTSD Knowledge | Day 0 baseline, 3 months
  Changes in levels of PTSD Knowledge measured by the PTSD Knowledge Test (0-14, higher scores indicating more PTSD knowledge).
Change in PTSD Related Stigma | Day 0 baseline, 3 months
  Changes in levels of PTSD Related Stigma measured by The Internalized Stigma of Mental Illness Scale (1 minimal stigma to 4 severe internalized stigma).
Change in Trauma-related cognitions | Day 0 baseline, 3 months
  Changes in levels of trauma-related cognitions assessed by the Post-Traumatic Cognitions Inventory (36-252 higher scores indicating higher incidence of negative trauma related cognitions).
Change in Self-reported arousal | Day 0 baseline, 3 months
  Changes in self-reported arousal levels measured with Self-Assessment Manikin (Self-Assessment Manikin measures arousal using 3 subscales: Valence, 1 unpleasant to 5 pleasant; Arousal rating, 1 calm to 5 excited; and Dominance, 1 independent to 5 dependent).
Change in Stress management strategy use | Day 0 baseline, 3 months
  Changes in use of the breathing retraining techniques as measured by self- and caregiver-reports during in-session homework review.
Change in Physiological arousal | Day 0 baseline, 3 months
  Changes in physiological arousal levels measured by heart rate variability (HRV).

SECONDARY OUTCOMES:
Change in PTSD Symptoms | Day 0 baseline, 3 months
  Changes in PTSD symptoms measured by the PTSD Checklist for Diagnostic Statistical Manual-5 (DSM-5; 0-80 higher scores indicating more severe symptoms).
Change in Depression Symptoms | Day 0 baseline, 3 months
  Changes in depression symptoms measured by the Patient Health Questionnaire (PHQ-9; 0-27 with higher scores indicating more severe depression).
Change in Anxiety Symptoms | Day 0 baseline, 3 months
  Changes in anxiety symptoms measured by the Generalized Anxiety Disorder-7 (GAD-7; 0-21 with higher scores indicating more severe anxiety).
Change in Functional impairment | Day 0 baseline, 3 months
  Changes in functional impairment assessed by the WHO Disability Assessment Schedule II (WHODAS 2.0; 0-48 with high scores indicating more severe functional impairment).

CONTACTS AND LOCATIONS:
Locations (1):
- Addis Ababa University, Addis Ababa, Ethiopia

REFERENCES:
- [Derived] Ng LC, Serba EG, Dubale BW, Fekadu A, Hanlon C. Posttraumatic stress disorder intervention for people with severe mental illness in a low-income country primary care setting: a randomized feasibility trial protocol. Pilot Feasibility Stud. 2021 Jul 30;7(1):149. doi: 10.1186/s40814-021-00883-3. PMID 34330334